CLINICAL TRIAL: NCT06379828
Title: Hospital Self-assessment Tool for the Implementation of the European Standards of Care for Newborn Health (ESCNH)
Brief Title: Self-assessment Tool for Implementing the ESCNH
Status: Not yet recruiting | Type: Observational
Sponsor: Global Foundation for the Care of Newborn Infants (Other)
Responsible Party: Principal Investigator, Luc Zimmermann, Senior Medical Director, Global Foundation for the Care of Newborn Infants
Other Study IDs: 2024-0140
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Development of a Tool to Assess the Level of Implementing the European Standards of Care for Newborn Health; Testing of the Developed Self-assessment Tool in European Hospitals; Self-Assessment
Keywords: ESCNH; EFCNI; eDlephi method; Pilot-testing; Implementation; Self-assessment; Tool; Neonatal care standards

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- eDelphi panel/participants: The eDelphi panels will consist of approximately 100 healthcare professionals from various European countries from the following fields: neonatology, midwifery, (neonatal) care, obstetrics, parent representing institutions, psychology, and physiotherapy. 20-30 of them will be invited for a final consensus workshop.
  Interventions: Other: Please note that this is an observational study; not applicable
- Pilot hospitals: 10 hospitals with neonatal units from Germany, UK, France, Italy, Sweden, Portugal, and Spain.
  Interventions: Other: Please note that this is an observational study; not applicable

INTERVENTIONS:
Other: Please note that this is an observational study; not applicable — Please note that this is an observational study; not applicable

SUMMARY:
This study aims to develop a tool for hospitals to self-assess the implementation of the European Standards of Care for Newborn Health (ESCNH), standards defining best-practice procedures for neonatal care. The tool shall support healthcare professionals across Europe to measure the level of implementation of the ESCNH, to identify variations in care delivery, and ultimately to improve neonatal care. To achieve this, healthcare professionals from all relevant backgrounds and parent representatives will be invited to take part in an electronic Delphi consensus approach. A subsequent pilot-testing among at least 10 hospitals across Europe will refine the developed tool, indicate potential errors, ensure user-friendliness, and improve the applicability.

DETAILED DESCRIPTION:
This project aims to develop a uniformly applicable self-assessment tool in different languages with the overall goal to support care providers across Europe to measure the level of implementation of the ESCNH, to pinpoint possible inhibitors, and ultimately to increase the extent of implementation. Covering the great variety of standards in one hands-on and easy-to-use self-assessment tool requires prioritising the most important components. This has to be approached in a systematic and scientific manner. For this purpose, a two-round electronic (e) Delphi survey will be conducted followed by an expert workshop. The aim of the two-stage eDelphi process is to lay a solid ground for the self-assessment tool. Prior to the eDelphi rounds, members of the study team together with the Project Expert Group (PEG) will condense and prioritise the ESCNH into one online questionnaire and thereby elaborate the first framework of the self-assessment tool. Next to participant-related information such as profession or country of employment, the questionnaire will cover specific aspects of the eleven major topics of the ESCNH namely: Birth and transfer, medical care and clinical practice, care procedures, infant- and family-centred developmental care, neonatal intensive care unit (NICU) design, nutrition, ethical decision-making and palliative care, follow-up and continuing care, patient safety and hygiene practice, data collection and documentation, education and training. The questionnaire will subsequently, in the first eDelphi round, be evaluated by the eDelphi panel. The panel consist of approximately 100 healthcare professionals from various disciplines related to neonatal care as well as parent representatives. In the first eDelphi round, panellists will appraise the relevance of included content, the wording of questions as well as the prioritisation of content to be included in the self-assessment tool. This will be enabled through a predefined evaluation scheme as well as free-text fields. Based on feedback from panellists, the preliminary self-assessment tool will be adapted by adding additional information, removing unnecessary items and re-wording if necessary. In the subsequent (second) eDelphi round, the same panellists will receive qualitative and quantitative information on the adaptation of the first version and will have again the option to evaluate the adapted questionnaire. Remaining discrepancies will be discussed in a final consensus workshop. For this purpose, 20-30 panellists will be selected based on their level of experience and invited for participation. The result of the workshop will be the agreed-upon content for the self-assessment tool. Except for the workshop, data collection during the eDelphi rounds will be anonymous.

To ensure applicability, the self-assessment tool will be pilot tested in European hospitals. For this purpose, the self-assessment tool will be translated into 5 languages (German, French, Italian, Swedish, Portuguese, and Spanish). For the pilot-testing, healthcare professionals in 10 pilot hospitals across Europe will be invited to evaluate the self-assessment tool. Feedback of the pilot-testing will be discussed with the PEG and adapted accordingly.

ELIGIBILITY:
Inclusion criteria Participants will be eligible if they are

* parent representatives or representatives of caregivers of infants who received special/intensive care,
* healthcare professionals in the field of neonatology, midwifery, neonatal nursing care, obstetrics, psychology, health sociology, physical therapy, or
* hospital management.

Exclusion Criteria Participants will be excluded if they

* provide insufficient proficiency of English for the eDelphi questionnaires or the languages of the self-assessment tool in the pilot testing, or
* have a professional background that is not related to the ESCNH / individuals that are not parent representatives or representatives of caregiver of infants who received special/intensive care.
* primarily work in the industry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The PEG consists of 8 renowned experts of multidisciplinary professions: neonatologists, a (neonatal) nurses, an obstetrician, a parent representative, a public health expert, and a statistician and is completed by members of the EFCNI study team.
  The eDelphi panels will consist of experts from various European countries from the following fields: neonatology, midwifery, (neonatal) care, obstetrics, parent representing institutions, psychology, and physiotherapy.
  Participants for the pilot-testing will be healthcare professionals with varying professional backgrounds in pilot hospitals across Europe.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-03 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Online self-assessment tool (including statements and questions) | 15.06.2024 - 15.07.2025
  Within a two-round eDelphi survey, the eDelphi panel will critically appraise the first template of the self-assessment tool. If required (indicated by ≥ 80% of participants) additional items will be added or unnecessary items will be removed. Remaining discrepancies will be discussed in a final consensus workshop and the questionnaire will be adapted based on consensus gathered within the workshop. The resulting questionnaire will be the first version of the self-assessment tool, which will be evaluated during and adapted after a pilot-testing phase.

SECONDARY OUTCOMES:
Response rates | 15.10.2024 - 30.06.2025
  Number of participants completing the first and second eDelphi round, number of hospitals joining the pilot-testing phase
Demographics and characteristics | 15.10.2024 - 30.06.2025
  A summary of demographic information and the participants characteristics will be presented
User-friendliness score of the self-assessment tool | 15.10.2024 - 30.06.2025
  Time taken to fill in, illustration on screen, understandability
Applicability score of the formulation of the questions | 15.10.2024 - 30.06.2025
  Evaluation data on formulation of the questions and understandability
Qualitative feedback on illustration of output | 15.10.2024 - 30.06.2025
  Evaluation data on illustration of questionnaire on the screen
Appraisal on the utilisation of the self-assessment tool | 15.10.2024 - 30.06.2025
  Evaluation data on the utilisation of the self-assessment tool
Scalability of the self-assessment tool and dissemination | 15.10.2024 - 30.06.2025
  Evaluation data on the usage and outreach

CONTACTS AND LOCATIONS:
Overall Officials: Silke Mader, Study Director — Global Foundation for the Care of Newborn Infants; Julia Hoffmann, Dr., Study Director — Global Foundation for the Care of Newborn Infants
Locations (1):
- European Foundation for the Care of Newborn Infants (EFCNI), Munich, Bavaria, Germany

REFERENCES:
- [Background] Lindacher V, Altebaeumer P, Marlow N, Matthaeus V, Straszewski IN, Thiele N, Pfeil JM, Zimmermann LJI, Mader S; European Standards of Care for Newborn Health project members. European Standards of Care for Newborn Health-A project protocol. Acta Paediatr. 2021 May;110(5):1433-1438. doi: 10.1111/apa.15712. Epub 2020 Dec 22. PMID 33290600
- [Derived] Hoffmann J, Lehmann S, Ancora G, Hummler H, Lack N, Schlembach D, Schouten E, Simonelli I, Thernstrom Blomqvist Y, Vavouraki E, Webbe J, Zimmermann LJI, Mader S, Geiger I. Study protocol for the development and pilot-testing of a Self-assessment tool for the implementation of the European Standards of Care for Newborn Health (ESCNH). BMJ Paediatr Open. 2025 Jan 20;9(1):e003008. doi: 10.1136/bmjpo-2024-003008. PMID 39837587
- See also: Related Info — https://newborn-health-standards.org/about/project-overview/
- Available data/document: Study Protocol — https://newborn-health-standards.org/about/project-overview/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/28/NCT06379828/Prot_SAP_000.pdf